CLINICAL TRIAL: NCT06739109
Title: Guided Internet-Based Treatment for Harmful Alcohol Use; EBehandling Alkohol
Acronym: eBA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset i Vestfold HF (Other)
Collaborators: Sykehuset Innlandet HF (Other); University Hospital, Akershus (Other); Hospital of Southern Norway Trust (Other); Trondheim University Hospital (Other)
Responsible Party: Principal Investigator, Kristin Klemmetsby Solli, Project leader, Sykehuset i Vestfold HF
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: eBehandling Alkohol; REK no 672168 (Other: REC south-east)
Record Dates: First submitted 2024-11-27; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Harmful Alcohol Use
Keywords: Internet based treatment; Guided internet treatment; Alcohol use
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- eBA intervention (Experimental): Adults with harmful alcohol use will be offered to complete a therapy-guided internet based intervention.
  Interventions: Procedure: Therapy-guided internet-based treatment program

INTERVENTIONS:
Procedure: Therapy-guided internet-based treatment program — eBA is a guided internet-based treatment for problematic alcohol use, based on cognitive behavioural therapy and motivational interview. The patients get access to self-help modules with information, questionnaires, and tools useful in a process of reducing alcohol use. Questionnaires measuring changes in alcohol use, illicit drug use, physical and mental health, and quality of life are frequently answered. These questionnaires are an integrated part of the treatment program and are used by the therapist to monitor and adjust the treatment according to each patient. The patients use the results from the questionnaires to assess whether the treatment is helpful reaching the treatment goal. The patients are guided by a therapist, and they communicate using a system for written messages in the treatment program and/ or guided by telephone.

SUMMARY:
Guided internet-based treatment for individuals with harmful alcohol use, eBehandling Alkohol (eBA), will be implemented as an experimental treatment option in five hospitals autumn 2024. Concurrently, a research project related to the effects of eBA will be conducted. Results from a pilot project show that treatment with eBA can help reduce alcohol use and improve mental health among people with harmful alcohol consumption. Similar results have been found in other international studies.

Many individuals with harmful alcohol consumption avoid seeking treatment, leading to negative consequences for the individual, their families, and society. The pilot project indicates that guided internet-based treatment is an effective treatment that is easily accessible and cost-effective. Access to eBA can help circumvent shame and stigma, increase access to treatment, reduce alcohol use, and improve physical and mental health.

Individuals who wish to participate in eBA do not need a referral from a GP. After an initial screening, participants will be given access to eBA, which consists of 9 treatment modules to be completed over an 8-12-week period, upon giving their consent. Participants will be followed up 4 weeks, 6 months, and 2 years after the completion of treatment. Data will be collected during screening, throughout the treatment period, and post-treatment. Data will be collected in the form of questionnaires, interviews, and registry data.

Simultaneously with the implementation of eBA as an experimental treatment, this project aims to investigate the characteristics of participants who apply for eBA, as well as examine the effects eBA may have in terms of reducing alcohol use, improving physical and mental health, and enhancing the quality of life among participants. The overarching goal of the study is to strengthen the understanding of the effects of internet-based treatment, thereby providing a sufficient basis to assess whether eBA should be implemented as a regular treatment option.

The study will also be part of a larger collaborative project where we will conduct meta-analyses of results from eBA and two other studies that also include treatment programs aimed at individuals with varying degrees of alcohol problems: the "Predictor Study" and "Endre". The three treatment programs are aimed at individuals who are at different stages in their problem trajectory. The goal of this collaborative project is to contribute to the development of a more holistic and targeted treatment offer for individuals with varying degrees of problem development.

DETAILED DESCRIPTION:
Introduction Harmful alcohol use is a pressing issue that affects individuals, families, and society as a whole, posing a significant public health problem. For the individual, harmful alcohol use can lead to mental and physical health issues, as well as social and relational problems. From a societal perspective, it can result in reduced work capacity, increased sickness absence, crime, violence, accidents, and injuries. In Norway, at least 17% of the adult population engages in potentially harmful alcohol consumption. This leads to many inpatient stays in both somatic and psychiatric hospitals. Reducing high alcohol consumption can yield substantial health benefits and significant societal savings.

The public health services for alcohol use disorder in Norway fall within the interdisciplinary specialized addiction treatment (Tverrfaglig Spesialisert Rusbehandling; TSB). TSB offers various treatment options, predominantly outpatient treatments through individual or group therapy sessions. An ongoing study at Vestfold Hospital Trust, titled "Patient factors predicting completion and outcome in group treatment of alcohol use disorders" (the "Predictor study"), explores how patient factors (psychological, sociodemographic, and societal) predict outcomes in group treatment for alcohol use disorders (AUD). This study tracks participants through approximately 3 months of treatment and follows up at 1 and 3 years post-treatment.

Despite available treatments, a significant proportion of people with emerging alcohol problems do not seek help early on, missing the opportunity for early intervention. The reasons for this reluctance are varied and complex. Feelings of shame and guilt over having an emerging alcohol problem can prevent some individuals from seeking health care. Additionally, treatment may be inaccessible, or the available treatment options may not be tailored to the individual's needs. Common barriers include the necessity for GP referrals for TSB treatments, the prioritization of treatment for severe cases of alcohol use, financial constraints, and the logistical challenges of traveling to outpatient clinics while balancing studies, work, or family responsibilities.

Needs Description eBA (eBehandling Alkohol) is a guided internet-based treatment for problematic alcohol use, developed through a collaboration between Vestfold Hospital Trust and Haukeland University Hospital. The treatment is grounded in cognitive behavioral therapy (CBT) and motivational interviewing (MI). It provides patients with access to self-help modules containing information, questionnaires, and tools useful for the process of reducing alcohol use. Patients regularly complete questionnaires that measure changes in alcohol use, other drug use, physical and mental health, and quality of life. These questionnaires are integrated into the treatment program and help therapists monitor and adjust the treatment. Patients can use their questionnaire results to assess whether the treatment is helping them achieve their goals. In the planned research project, data from these questionnaires will be utilized to answer the research questions. Patients are guided by therapists through written messages in the treatment program or by telephone.

One of the main advantages of eBA is the potential to offer treatment for harmful alcohol use at an early stage, thus preventing further deterioration of the problem. This is invaluable for individuals, their families, and society. eBA is easily accessible, discrete, and can lower the threshold for seeking help by reducing stigma, financial barriers, and logistical difficulties.

Evidence from a pilot study using participant data from eBA showed promising results. The participants had a mean age of 49 years, with 60% being men, 65% having a partner, and 76% having children. Approximately 75% of the participants reported a reduction in alcohol use, and reported reduced symptoms of anxiety and depression. These results align with international research that supports guided internet-based treatment for emerging alcohol problems as an effective means of reducing alcohol use and improving mental health. Other studies have shown similar treatments to be helpful for a range of addiction-related problems. However, despite this research, internet-based treatment for alcohol misuse has not yet been broadly implemented in health services.

Project Methodology The proposed study will be a prospective multicentre cohort study, following individuals with harmful alcohol use from the initial screening interview, through the start of treatment, during the 9 treatment modules, and at follow-ups at 1 month, 6 months, and 2 years after treatment completion.

The target group for this project comprises adult men and women with problematic alcohol use who, for various reasons, do not seek help through traditional treatment options. These individuals must be willing to make an effort to reduce their alcohol use and be eligible to use guided internet-based treatment. Participants must have access to a computer, tablet, or smartphone and be able to securely access the internet-based treatment using BankID. Recruitment will be conducted through press releases, social media, and leaflets distributed at outpatient clinics and GP offices. Interested individuals can inquire about participation by sending an SMS. A therapist will then contact the participants for an initial interview. Inclusion in the study will be based on written informed consent and meeting the inclusion criteria.

The questionnaires used in this study are mainly equivalent to those implemented in other guided internet-based treatment programs in Norway, allowing for comparative analysis. Post-treatment efficacy will be assessed at 1 month, 6 months, and 2 years post-treatment. The questionnaires will cover various domains, including demographics, age, sex, education, occupation, main source of income, marital status, children, duration of the problem, previous treatment experience, patient goals, planned alcohol use, drinking patterns, daily alcohol consumption, AUDIT (Alcohol Use Disorder Scale), DUDIT (Drug User Disorder Scale), PHQ-9 (Patient Health Questionnaire), GAD-7 (Generalized Anxiety Disorder), 5Q-5D-5L + VAS (quality of life and treatment satisfaction), DTCQ (Drug Taking Confidence Questionnaire), SCL-10R (Symptom Check List), C-scale (User satisfaction), WHO-1 quality of life, and evaluation & goal achievement.

Participants will also consent to the collection of registry data for 1 year prior to treatment start and 2 years after treatment completion. Information about the type and amount of treatment received from specialized and municipal health services will be collected through databases from the Norwegian Patient Registry, the Control and Payment of Health Refunds Registry, and causes of death from the Cause of Death Registry. Qualitative interviews will be conducted through individual semi-structured interviews with approximately 20 participants who specifically consent to this interview.

The Predictor study and the Endre study are collecting data that overlap with the eBA study in several areas, providing a basis for conducting meta-analyses. Data compared from the three studies will be anonymized and aggregated at the group level.

The pilot study indicated an average decrease in AUDIT score from pre-treatment to module 8 (T2) of 3.45, with a standard deviation of 4.76. With a sample size of 250 individuals, the width of a 95% confidence interval is estimated at 1.23, with a probability of 0.8 of achieving the estimated width. This interval width increases to 1.55 if the final sample size at module 8 is reduced to 160 individuals due to a 36% dropout. Adjusting for additional factors in the statistical analysis requires an increase in sample size. Given these precision estimates, accounting for potential dropouts, and the need to adjust for additional factors, a sample size of 250 individuals is satisfactory.

Treatment outcome/retention in treatment will be analyzed using survival analyses such as Kaplan-Meier/Cox regression. Outcome measures will undergo regression analyses on short-term (T2) and long-term (T4 and T5) outcomes, with primary measures being alcohol use, physical and mental health symptoms, and quality of life. Descriptive data will be provided as mean and/or median values, along with standard deviations and/or 95% confidence intervals. The significance level/p value is set to < 0.05. Meta-analyses will be conducted using data from the eBA study, the Predictor study, and the Endre study.

Participants, Organization, and Collaborations The eBA program and the associated study will be managed and organized from Vestfold Hospital Trust. The Division of Mental Health and Addiction was responsible for developing eBA as an experimental treatment program and for conducting the pilot study. This division has expertise at all levels of implementing and conducting guided internet-treatment programs. Several hospitals will participate in eBA implementation: Sørlandet Hospital Trust, Akershus University Hospital, Innlandet Hospital Trust, St. Olavs Hospital, and Vestfold Hospital Trust. Written agreements will ensure cooperation among these hospitals. A project group will be established to coordinate the daily operations of the treatment program. This group will comprise local representatives from Vestfold Hospital Trust and coordinators at the collaborating institutions. Designated clinicians at participating hospitals will receive training and supervision from experienced clinicians at Vestfold Hospital Trust. A steering committee for the research project will include representatives from the participating hospitals and the Predictor and Endre studies, as well as a user representative. The Research Group for Substance Use and Addiction at Vestfold Hospital Trust will serve as the reference group for the research project.For research independence, researchers and the PhD candidate will not perform tasks involving therapeutic guidance of participants.

Plan for Implementation eBA, trialed as an experimental treatment at Vestfold Hospital Trust, will be implemented as a treatment option in selected hospitals in 2024. The questionnaires integrated into the eBA program assessing alcohol use, somatic, and mental health will enable seamless data collection for the research project. The study's results will inform whether eBA can become a standard treatment option for people with harmful alcohol use. The goal is to demonstrate positive outcomes and satisfaction, highlighting eBA's accessibility, potential to increase treatment numbers, and cost-effectiveness. Findings will be shared with health authorities and published in high-ranking international peer-reviewed journals.

Given its close link to clinical practice, the research results will be readily relevant for clinicians. The implementation of eBA is expected to utilize existing resources within Norway's substance use disorder treatment infrastructure. Clinicians are familiar with this patient group and their follow-up needs.

A meta-analysis comparing results from eBA, the Predictor study, and the Endre study is anticipated to clarify which individuals benefit most from different treatment options. Offering varied treatments tailored to each individual's stage of problem development is crucial for providing comprehensive care.

User Involvement The Addiction Research Group at Vestfold Hospital Trust, including a user representative, will act as the project's reference group. The user representative has been involved in drafting the project outline and research questions and will continue to advise on and participate in the study throughout its duration.

Ethical Considerations Adhering to the Helsinki Declaration's principles and other applicable regulatory requirements, the study will maintain high ethical standards. Participants' data will be registered per national personal data laws, with approval from regional ethical committees and Data Protection Officers at each participating hospital. To safeguard research independence, the researchers or PhD candidate will not conduct tasks involving therapeutic guidance of participants.

Participants will provide written consent before inclusion and can withdraw at any time. Recruitment will include both genders, and any significant gender-focused findings will be reported. The study does not involve environmental concerns. Clinicians will monitor participants throughout the project and refer them to traditional treatments if needed.

By thoroughly documenting the structured assessment, implementation, and potential broader adoption of eBA, this detailed project framework aims to reduce harmful alcohol use through innovative internet-based treatments. These treatments are anticipated to be effective, accessible, and broadly beneficial, offering significant improvements in public health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Harmful alcohol use
* Willing to make an effort to reduce alcohol consumption
* Able to use guided internet-based treatment
* Access to a computer, tablet, or smartphone
* Access to BankID or equivalent secure log-in

Exclusion Criteria:

* Acute and/or severe mental disorders, such as psychotic issues or ongoing suicidal issues.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Identifying characteristics of people seeking eBA | Baseline measure
  Describe demographics, age, sex, education, occupation, main source of income, marital status, children, duration of problem, previous treatment experience
Changes in alcohol use | Measure changes from baseline to end of treatment, and 6 months and 2 years post-treatment
  Measure changes using the Alcohol Use Disorder Scale (AUDIT ), reporting on a sum score scale from 0 to 40; higher score indicate worse outcome.
Changes in mental health status | Measure changes from baseline to end of treatment, and 6 months and 2 years post-treatment
  Measure changes in SCL-10R (Symptom Check List) scores on a scale from 1 to 4, the higher score the wore outcome.
Changes in mental health status | Measure changes from baseline to end of treatment, and 6 months and 2 years post-treatment
  Measure changes using GAD-7 (Generalized Anxiety Disorder), reporting on a scale from 0 to 3; higher score indicating worse outcome.
Changes in quality of life | Measure changes from baseline to end of treatment, and 6 months and 2 years post-treatment
  Measure changes in 5Q-5D-5L (quality of life ), including av visual analoge scale (VAS). The 5Q-5D-5L scores on a scale from 1 to 5, were high score indicate worse outcome. The instrument includes a VAS from 0 to 100, where higher score indicate better outcome.
Changes in quality of life | Measure changes from baseline to end of treatment, and 6 months and 2 years post-treatment
  Measure changes in WHO quality of life score (WHOQOL-1) on a scale from 1 to 5, where higher scores indicate better outcome.

SECONDARY OUTCOMES:
Compare participants characteristics in the eBA study, the Predictor Study and the Endre study | Baseline measure
  Compare distribuation of gender, age and The Alcohol Use Disorder Scale (AUDIT) scores between the 3 studies. AUDIT reports on a sum score scale from 0 to 40; higher score indicate worse outcome.
Compare retention in treatment in eBA to standard group-treatment in the Predictor study and the Endre program | End of treatment program
  Number of participants completing the 3 studies.
Compare changes in alcohol use between participants in the eBA study, the Predictor study and the Endre study | Measure changes from baseline to end of treatment, and 6 months and 2 years post-treatment
  Compare changes in The Alcohol Use Disorder Scale (AUDIT ) scores between the 3 studies. AUDIT reports on a sum score scale from 0 to 40; higher score indicate worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin K Solli, PhD, Principal Investigator — Sykehuset i Vestfold HF
Locations (5):
- Norway (5):
  - Sørlandet Hospital Trust (Hospital of Kristiansand), Kristiansand, Agder
  - Akershus University Hospital, Loerenskog, Akershus
  - Innlandet Hospital Trust, Lillehammer, Innlandet
  - St. Olavs Hospital, Trondheim, Trøndelag
  - Vestfold Hospital Trust, Tønsberg, Vestfold

IPD SHARING:
Plan to Share IPD: No
With the aim of doing a meta analysis, we will share anonymized aggregated data at the group level with the research leaders of the Predictor study and the Endre study. In consideration of the participating patients' rights, we will not share individual participant data.

REFERENCES:
- See also: Information about the eBA intervention in the Web sites of Vestfold Hospital Trust — https://www.siv.no/ebehandling/ebehandling-alkohol/